CLINICAL TRIAL: NCT03757273
Title: Aesthetic Reconstruction of Onco-surgical Mandibular Defects Using Free Fibular Flap With and Without CAD/CAM Customized Osteotomy Guide (A Randomized Controlled Clinical Trial)
Brief Title: Aesthetic Reconstruction of Onco-surgical Mandibular Defects Using FFF With and Without CAD/CAM Customized Cutting Guide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Esmail Abdullah Al-Sabahi, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 653
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Mandibular Tumors
Keywords: Mandibular tumors resection/reconstruction; CAD/CAM; Osteotomy, Cutting guide; Aesthetic; Operation time; Free fibular flap

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Because the two interventions used in this trial are easily recognized by the participant and the investigators, neither the investigator nor the participant can be blinded. But, the assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FFF with CAD/CAM customized cutting guide (Experimental): Mandibular reconstruction using free fibular flap with CAD/CAM customized osteotomy guide.
  Interventions: Procedure: FFF with CAD/CAM customized cutting guide
- FFF without customized cutting guide (Active Comparator): Mandibular reconstruction using free fibular flap without customized osteotomy guide. CAD/CAM 3D model for mandible will be used.
  Interventions: Procedure: FFF without customized cutting guide

INTERVENTIONS:
Procedure: FFF with CAD/CAM customized cutting guide — This began with the acquisition of a high-resolution CT scan of the craniofacial skeleton and lower legs. the CT scan will be sent to the modeling company for producing autoclavable 3D models and cutting guides of the mandible and fibula to be used during the workflow as well as a model of the final reconstructed mandible. Surgery will be performed by two surgical teams, one for cervicofacial resection and the other harvesting the flap. access to the mandible is obtained, osteotomy guides secured; cuts then accomplished as planned virtually. fibular flap is harvested and cutting guides secured to replicate osteotomies and reshaping as planned to conform with remaining mandible. fixation and pedicle anastomosis is performed. Finally, the operation completed with soft tissue reconstruction.
  Arms: FFF with CAD/CAM customized cutting guide
Procedure: FFF without customized cutting guide — This began with the acquisition of a high-resolution CT scan of the craniofacial skeleton. the C.T scan will be sent to the modeling company for planning three-dimensional model of the mandible. autoclavable model will be prepared for mandible to be used during the workflow for plate reshaping and positioning to conform with the remaining mandible.
  Surgery will be performed by two surgical teams, one in charge of cervicofacial resection and the other harvesting the flap. access to the mandible is obtained, and resection/ reconstruction then performed in conventional surgical manner with microvascular anastomosis. Finally, the operation will be completed with soft tissue reconstruction.
  Arms: FFF without customized cutting guide

SUMMARY:
The purpose of this study is to compare Aesthetic results and operation time of free fibular flap with and without CAD/CAM customized osteotomy guide for reconstruction of mandibular defects.

DETAILED DESCRIPTION:
Oral and maxillofacial tumors posing an important fact as a demanding challenge for surgeons causing face disfigurement which require post-ablation reconstruction. One of the most challenging procedure facing reconstructive surgeons lies in mandibular defects after tumor resection causing facial disharmony affecting aesthetics and function.

Free flaps are considered the gold standard for the reconstruction during oncologic surgery combining a high success rate with low donor site morbidity. Various techniques have been practiced and performed in mandibular defect reconstruction. Hidalgo introduced the fibular graft as an option, offering many Assorted advantages: as it provides a sufficient source for bone and soft tissue harvesting; long reliable vascular pedicle; moreover, only minor donor site morbidity may be involved and flap harvesting require no patient reposition.

Mandibular reconstruction using FFF has become the gold standard. However, flap contouring remain an issue and imprecise with inconvenient or suboptimal final results regrading aesthetic and even more consuming time and efforts owing to poor planning when performed traditionally. Recently, with newly introduced technology and virtual planning, the process has become more uniform and reproducible thus enhancing final outcome improving patient life.

Prefabricated cutting guides may be used may be not, however it still in debate regarding its benefits and worth for patient and surgeon. believing that ability of CAD/CAM technology to achieve Aesthetic and operation time improvement with more detailed evaluation in patients undergoing mandibular reconstruction using free fibular flap with CAD/CAM customized cutting guide.

Our priori-hypothesis is that utilization of CAD/CAM-assisted with customized osteotomy guide is not related to an altered result regarding aesthetic outcome and operation time in patient undergoing mandibular reconstruction using free fibular flap. In order to test this hypothesis, we will compare aesthetic outcome and operation time in group of patients receive FFF by CAD/CAM-assisted with customized osteotomy guide to the results of another group of patients receive FFF but without customized osteotomy guide. only model will be performed as conventional method helping in pre-shaping of reconstruction plate which is another well-established concept of management of mandibular defect.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by tumor involving Mandibular bone.

Exclusion Criteria:

* Patients having poor oncological prognosis
* Patients with poor performance status together with other relative or absolute vascular contraindication.
* Patients require marginal resection or with bilateral fibular fracture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Aesthetic | at least three months post operative
  Aesthetic outcome will be measured objectively by computerized digital analysis as differential angle and differential area of reconstructed to the other side of the mandible. subjectively will be evaluated using VAS.

SECONDARY OUTCOMES:
Operation time | intraoperative
  Operation time will be recorded intraoperatively in the surgery day as total operation time and ischemia time.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Al-Sabahi, Phd. student, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Sabahi ME, Jamali OM, Shindy MI, Moussa BG, Amin AA, Zedan MH. Aesthetic Reconstruction of Onco-surgical Mandibular Defects Using Free Fibular Flap with and without CAD/CAM Customized Osteotomy Guide: A Randomized Controlled Clinical Trial. BMC Cancer. 2022 Dec 2;22(1):1252. doi: 10.1186/s12885-022-10322-y. PMID 36460978